CLINICAL TRIAL: NCT04797689
Title: Managing Our Relationship With Food and Eating
Acronym: NOURISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lethbridge (Other)
Responsible Party: Principal Investigator, Cheryl Currie, Associate Professor, University of Lethbridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021 - 020
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Mental Health Wellness 1; Eating Behavior; Stress, Psychological; Eating Habit
MeSH Terms: conditions — Feeding Behavior; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trauma Informed Yoga (Experimental): Participants will receive 12 x 60 min group-based yoga sessions, delivered synchronously over Zoom.
  Interventions: Behavioral: Trauma Informed Yoga
- Trauma Informed Psychotherapy (Experimental): Participants will receive 12 x 120 min group-based psychotherapy sessions, delivered synchronously over Zoom.
  Interventions: Behavioral: Trauma Informed Psychotherapy
- Control (No Intervention): These participants will not receive an intervention.

INTERVENTIONS:
Behavioral: Trauma Informed Yoga — One licensed yoga instructor, trained in trauma-informed yoga delivery, will lead the online sessions. Participants will be instructed to engage in the class from a mat or chair in their home or move between them as the class unfolds. The instructor will begin the class by introducing the week's theme (e.g. grounding and safety, non-attachment, imprints of the past and impacts on our reactions to COVID-19, connection to nature), followed by a breath practice (10 min), a yoga practice (50 min), a meditation practice (10 min), and closing words (10 min).
  Arms: Trauma Informed Yoga
Behavioral: Trauma Informed Psychotherapy — Two licensed counsellors (MSW-trained) will co-facilitate the online version of this program. Facilitators will begin the session by introducing the week's theme (e.g. setting goals while working from home, being mindful, health coping) (10 min), followed by a lecture and activity to integrate learning (e.g. large and small group discussion using Zoom break out rooms, journaling) (70 min), and closing words (10 min).
  Arms: Trauma Informed Psychotherapy

SUMMARY:
There is a need for population-level intervention research to address the impacts of the COVID-19 pandemic on disordered eating and unhealthy eating behaviours. Systematic reviews have demonstrated that psychotherapy and yoga can help to reduce binge eating and disordered eating habits, however, these interventions were tested in person. Studies examining the effectiveness of these interventions in an online, group-based format are warranted. In 2019, the investigators launched a RCT to test gender-stratified group interventions to address mental health and addictive behaviours among community-based adults in southern Alberta. The investigators implemented this intervention with more than 200 adults in person before this study was paused due to COVID-19; In 2020, the investigators adapted this intervention for online delivery to 200 community-dwelling women across Alberta. The most recent iteration of this study indicated the participants were particularly concerned about their relationship with food and how they were engaging in different eating behaviours to cope with the stress of COVID-19.

DETAILED DESCRIPTION:
The primary objective of this project is to adapt two existing mental health and substance use interventions and RCT for online delivery to address unhealthy eating behaviours and a negative relationship with food for women within the context of COVID-19. The second objective is to test if an online group body-oriented intervention (trauma-sensitive yoga) that has been designed to increase awareness of physical sensations, is superior to an online group verbal narrative intervention (mental wellness talking circle), and to control group. The investigators theorize that the body-oriented intervention may offer the opportunity to reprogram automatic physiologic hyperarousal in response to COVID-19 triggers and increase positive body awareness, and mindful attention to the ways in which habitual self-protective behaviours, like unhealthy eating behaviours, may be impacting health. The third objective is to examine the impacts of the interventions on adults with pre-existing mental health and disordered eating issues, and those with previous experiences that may make them more susceptible to these problems during COVID-19. The investigators will track other supports they engage in during the study and the perceived impacts of these supports on their outcomes with the goal of shedding light on how to best match COVID-19 related services to adults who need them the most.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-75 years living in Alberta, Canada
* Need to have reliable access to the internet, a device with a webcam for the next 2 months
* Need to self-identify that they are currently struggling with at least one of: stress eating, alcohol use, drug use, tobacco use, or gambling during the pandemic

Exclusion Criteria:

* Non-community dwelling
* Not currently residing in Alberta, Canada

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Changes in Intuitive Eating Behaviours | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Intuitive eating behaviours will be assessed using the 23-item The Intuitive Eating Scale-2 (IES-2). Items are measured on a 5-point Likert, with options ranging from "Strongly Disagree" to "Strongly Agree". Among women, the IES-2 has good internal consistency (α = 0.87), good convergent validity with the original IES (r = 0.87), and strong test-retest reliability (r = 0.88).

SECONDARY OUTCOMES:
Changes in Anxiety and Depression | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Anxiety and depression will be assessed through the 14-item Hospital Anxiety and Depression Scale (HADS). Seven items assess anxiety while the remaining seven measure depression. There are four response options (0-3), which create scale values from 0-21 for each scale. Three ranges of scores have been identified: 0-7 (non-cases), 8-10 (doubtful cases) and 11-21 (cases).
Changes in addictive eating behaviours | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  To assess addiction-like eating behaviours, questions regarding food cravings, loss of control over food and eating, prioritization of food and eating, and guilty feelings due to food or eating will be measured on a 5-point Likert scale with frequencies ranging from "Never" to "4+ times per week". Questions regarding concern from others will be measured on a 3-point Likert scale, with the options "Never", "Yes, but not in the past year", and "Yes, in the past year".

OTHER OUTCOMES:
Changes in Body Image | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  The 12-item Body Image-Acceptance and Action Questionnaire (BI-AAQ) will be used to assess participants' flexibility with their body image. The items are measured on a 7-point Likert scale, with options ranging from "Never True" to "Always True". The BI-AAQ has excellent internal consistency across three samples (α range = 0.92 - 0.93), good test-retest reliability (r = 0.80), and showed divergent validity with body image dissatisfaction (r = -0.80), dieting (r = -0.70), food preoccupation (r = -0.61), and oral control (r = -0.27).
Changes in Internalized Weight Bias | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Participant experience with weight-based self-stigma will be assessed using 10 items of the 11-item Modified Weight Bias Internalization Scale (WBIS-M). Items are measured on a 7-point Likert scale with options ranging from "Strongly Disagree" to "Strongly Agree". The WBIS-M has excellent internal consistency (α = 0.94), and is valid against relevant psychological measures. The WBIS-M will be administered at all timepoints to assess changes in weight-based self-stigma over the intervention period.
Changes in Tobacco Use | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Participants will be asked to self-report if tobacco use has changed during the pandemic via a 5-point likert. Options range from increased a lot to decreased a lot. If participants indicate their tobacco use has changed, they will be asked to identify the primary reason for this change. Changes in tobacco use will be re-assessed at each time point.
Changes in Alcohol Use | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Past year alcohol consumption will be assessed through the Alcohol Use Disorder Identification Test (AUDIT). Scores on the AUDIT range from 0 to 40; a score over 8 is indicative of problematic or hazardous alcohol use. Changes in alcohol consumption since the beginning of the pandemic will be identified through a 5-point likert. Changes in alcohol use will be re-assessed at each time point.
Changes in Cannabis Use | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Past year cannabis use will be assessed through the Cannabis Use Disorder Identification Test - Revised. Scores range from 0-31; a score over 8 is indicative of problematic or hazardous use. Changes in cannabis use will be re-assessed at each time point.
Changes in Physical Activity and Sedentary Behaviour | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Physical activity will be assessed through the International Physical Activity Questionnaire - Short Form. The questionnaire asks about frequency and duration of vigorous (VPA) and moderate physical activity (MPA) over the past 7 days. Weekly Metabolic Equivalents (MET) minutes will be calculated based on responses. Participants will be categorized into high (>1500 MET min/week with 3+ days of VPA or >3000 METmin/week with 7+ days of MVPA); medium (5+ days of 20+ minutes of VPA per day, 5+ days with 30+ minutes of MPA per day, or 5+ days of MVPA that achieves 600+ MET min/week); low (participant does not meet other cut points). Frequency and duration of walking and sitting time are also assessed. The IPAQ has good reliability and criterion validity.
Changes in Self-Esteem | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Self-esteem will be measured using the 10-item Rosenberg Self Esteem Scale. The scale is a widely used measure that correlates well with other measures of self-esteem and has strong internal consistency (0.92) and test-retest reliability (0.88). Scores range from 4 to 40; a higher score indicates higher self esteem.
Changes in Loneliness | Baseline, Mid-point (6 weeks), Post-Intervention (12 weeks)
  Loneliness will be evaluated using a shortened (3 item) version of the UCLA Loneliness Scale. This scale asks about feelings of companionship, being left out, and being isolated from others in the last month, with a 3-item list of answer options (hardly ever, some of the time, often). This scale has good reliability (r = 0.73), validity, and internal consistency (Cronbach's α = 0.84-0.94). The scale also showed convergent validity with other commonly used measures of loneliness. Scores range from 1 to 9; higher scores indicate higher levels of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Currie, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- University of Lethbridge, Lethbridge, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data relevant to the researcher's research question may be shared upon a reasonable request
Time Frame: January 2023, for up to 10 years
Access Criteria: Researchers must make a reasonable request to the PI